CLINICAL TRIAL: NCT04487015
Title: Digital Approaches to Improve Carbohydrate Periodisation Behaviour in Athletes Using a Pilot Sequential Multiple Assignment Randomised Trial Design.
Brief Title: A Digital Approach to Improving Carbohydrate Periodisation Behaviours in Athlete: SMART+ Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Liverpool John Moores University (Other)
Collaborators: Applied Behaviour Systems Ltd (Unknown); University College, London (Other); Duke-NUS Graduate Medical School (Other)
Responsible Party: Principal Investigator, David Dunne, PhD Student, Liverpool John Moores University
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: 20/NSP/027
Record Dates: First submitted 2020-07-22; First posted 2020-07-27 (Actual); Last update posted 2020-11-27 (Actual); Status verified 2020-11

CONDITIONS: Diet Habit
Keywords: carbohydrate periodisation; mobile app; nutrition; adaptive design; behaviour change; digital intervention; sports performance; technology
MeSH Terms: conditions — Feeding Behavior | interventions — CD56 Antigen

STUDY DESIGN:
Intervention Model Description: Sequential Multiple Assignment Randomized Trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (9):
- Part I: Non-Digital (Control) (No Intervention): Participants who currently receive performance nutrition support, via a qualified practitioner as indicated by a member of the sports science team at their sporting organisation, will be assigned to the non-digital approach (control). These participants will not receive any intervention from the research team for the duration of this study (6 weeks).
- Part I: MP+ Call + MesC [6 weeks] (Experimental): For part one of study, participants who currently do not receive performance nutrition support, will be given access to an app-based menu planner (MP) for 6 weeks with coach support that gives ad-hoc messaging and calls.
  Interventions: Behavioral: MP; Behavioral: Call; Behavioral: MesC
- Part II: Stage 1- MP [1week] (Experimental): For the pilot SMART trial (part two of study), participants (not the same participants as part one) who currently do not receive performance nutrition support, will be given access to a menu planner app (MP) for 4 weeks. In the first 1 week, participants will only receive MP.
  Interventions: Behavioral: MP
- Part II: Stage 2 - R1-MP [1 week] (Experimental): For participants in Part II: Stage 1- MP [1week], after the first 1week, this group of participants are considered responders (R1) so they continue with MP only for another 1 week.
  Participants' response status is dependent on whether they are randomised to using the stringent or relaxed engagement criteria as described in study details.
  Interventions: Behavioral: MP
- Part II: Stage 2 - NR1-MP [1 week] (Experimental): For participants in Part II: Stage 1- MP [1week], after the first 1 week, this group of participants are considered non-responders (NR1) and are re-randomised to continue with MP only for another 1 week.
  Participants' response status is dependent on whether they are randomised to using the stringent or relaxed engagement criteria as described in study details.
  Interventions: Behavioral: MP
- Part II: Stage 2 - NR1-MP + Call + MesC [1 week] (Experimental): For participants in Part II: Stage 1- MP [1 week], after the first 1 week, this group of participants are considered non-responders (NR1) and are re-randomised to have MP and additional coach support for another 1 week. The coach support consists of up to 3 coach-initiated messaging and ad-hoc calls to participant.
  Participants' response status is dependent on whether they are randomised to using the stringent or relaxed engagement criteria as described in study details.
  Interventions: Behavioral: MP; Behavioral: Call; Behavioral: MesC
- Part II: Stage 3 - R2-MP [2 weeks] (Experimental): After going through Part II: Stage 2, this group of participants are considered responders (R2) so they continue with MP only for 2 weeks.
  Participants' response status is dependent on whether they are randomised to using the stringent or relaxed engagement criteria as described in study details.
  Interventions: Behavioral: MP
- Part II: Stage 3 - NR2-MP [2 weeks] (Experimental): After going through Part II: Stage 2, this group of participants are considered non-responders (NR2) and are re-randomised to use MP only for another 2 week.
  Participants' response status is dependent on whether they are randomised to using the stringent or relaxed engagement criteria as described in study details.
  Interventions: Behavioral: MP
- Part II: Stage 3 - NR2-MP + Call + MesC [2 weeks] (Experimental): After going through Part II: Stage 2, this group of participants are considered non-responders (NR2) and are re-randomised to have MP and additional coach support for another 2 weeks. The coach support consists of up to 3 coach-initiated messaging and ad-hoc calls to participant.
  Participants' response status is dependent on whether they are randomised to using the stringent or relaxed engagement criteria as described in study details.
  Interventions: Behavioral: MP; Behavioral: Call; Behavioral: MesC

INTERVENTIONS:
Behavioral: MP — The app-based menu planner (MP) given to the participants has an automated carbohydrate periodisation menu planning tool, an educational and motivational nutrition content (infographics, video and text articles), and recipes. Participants using the app will input their training schedule into the app to produce their own menu plans. The behaviour change techniques (BCT) underlying the intervention are goal & planning, feedback & monitoring, shaping knowledge, natural consequences, comparison of behaviour, comparison of outcome, associations, repetitions, reward & threat, regulation and antecedents.
  Arms: Part I: MP+ Call + MesC [6 weeks]; Part II: Stage 1- MP [1week]; Part II: Stage 2 - NR1-MP + Call + MesC [1 week]; Part II: Stage 2 - NR1-MP [1 week]; Part II: Stage 2 - R1-MP [1 week]; Part II: Stage 3 - NR2-MP + Call + MesC [2 weeks]; Part II: Stage 3 - NR2-MP [2 weeks]; Part II: Stage 3 - R2-MP [2 weeks]
Behavioral: Call — A 30-45 minutes coaching consultation telephone/Skype call from the nutrition coaching to give social support. The BCT underlying the intervention is goal & planning, social support, natural consequences.
  Arms: Part I: MP+ Call + MesC [6 weeks]; Part II: Stage 2 - NR1-MP + Call + MesC [1 week]; Part II: Stage 3 - NR2-MP + Call + MesC [2 weeks]
Behavioral: MesC — Nutrition coach-led messaging (MesC) is where the mobile app (MP) has the text messaging feature activated, and the nutrition coach proactively initiates a conversation via text messaging up to three times a week to offer nutrition support to the participant. The BCT underlying the intervention is goal & planning, social support, natural consequences.
  Arms: Part I: MP+ Call + MesC [6 weeks]; Part II: Stage 2 - NR1-MP + Call + MesC [1 week]; Part II: Stage 3 - NR2-MP + Call + MesC [2 weeks]

SUMMARY:
The carbohydrate periodisation framework is a widely accepted nutritional intervention strategy in the field of sports nutrition. However, despite the validity of this approach, it is reported that athletes find it difficult to stick to this behaviour and that the support required is highly personalised, and as a result time consuming for the coach. Prior research has suggested that a digital environment can deliver better personalised dietary interventions to better support athletes.

The overall purpose of this study is to assess the feasibility and acceptability of a digital approach (a menu planner app with coach support), and gain understanding on the strategy to implement coach support according to app engagement in the digital approach to improve dietary carbohydrate periodisation behaviours in athletes.

DETAILED DESCRIPTION:
The study is conducted in two consecutive parts.

For part one, to assess the feasibility and acceptability of the digital approach, participants are recruited to use the app for 6 weeks and were given coach support, where coaches message (MesC) and call (ad-hoc Call) and the participants. A control group (no app) is also separately recruited to compare with the menu planner group.

For part two, to gain better understanding on the strategy to implement coach support with the menu planner app according to app engagement, a pilot multiple assignment randomized trial (SMART) design is conducted. Participants are equally randomised to either receive a stringent engagement criteria strategy or relaxed adherence criteria strategy. A stringent engagement criteria strategy requires the user to use the app at least twice a week at stage 1, and at least 3 times a week at stage 2 to be considered a responder at stage 1 and stage 2 (R1 and R2).

A relaxed engagement criteria strategy requires the user to use the app at least once a week in week 1 of using the app at stage 1, and at least 2 times a week at stage 2, to be considered a responder at stage 1 and stage 2 (R1 and R2). Non-responders for both criteria strategies at stage 1 and 2 (NR1 and NR2) will be re-randomised to either continue with the app only or additional coach support (MesC + ad-hoc Call).

Timeline wise,

Stage 1: Participants will first receive app for 1 week and will be categorised as responder (R1) or non-responders (NR1) at the end of the 1 week.

Stage 2: Responders to stage 1 (R1) will continue with the menu planner for 1 week. Non-responders to stage 1 (NR1) will either continue with the menu planner or receive additional coach support (MesC + ad-hoc Call) for 1 week. Participants are categorised again as responder (R2) or non-responders (NR2) at the end of the week.

Stage 3: Responders to stage 2 (R2) will only have menu planner for 2 weeks. Non-responders to stage 2 (NR2) will either have menu planner only or receive/continue with additional coach support (MesC + ad-hoc Call) for 2 weeks.

The SMART trial will take a total of 4 weeks to complete and have up to two randomisation points per participant. All re-randomisations are done at 1:1 allocation ratio.

ELIGIBILITY:
Inclusion Criteria:

* Have access to a personal smart phone.
* An elite or training athlete.
* Have a performance related weight loss or weight maintenance physical goal.
* Do not have or have not have a history of eating disorders or disordered eating.

Exclusion Criteria:

* Participants with a medically diagnosed history of eating disorders or disordered eating will be asked to self-exclude from the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1000 (Estimated)
Dates: Start 2020-09-14 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Success rates of carbohydrate periodisation behaviour at week 4, 6 | At week 6 (for part I of study) and week 4 (part II of study)
  A binary success of whether dietary periodisation behaviour has improved in the participant measured by the "periodisation behaviour questionnaire" (in the process of submitting the paper on validation of questionnaire). The scale is 1- does not periodise, 2-periodises energy but not carbohydrate, and 3-periodises both. Higher score indicates better periodisation behaviour. Only score of 3 is considered success.

SECONDARY OUTCOMES:
Change in dietary self-efficacy from baseline to week 4, 6 | At baseline (week 0) and at week 6 (for part I of study) and week 4 (part II of study)
  The dietary self-efficacy will be assessed using a self-efficacy scale. This questionnaire have been validated in the general population (Stich, Knauper and Tint, 2009). The scale is a 5-point scale from 1 for not confident at all, to 5 for very confident. Higher score indicates higher self-efficacy.
Change in beliefs about consequences from baseline to week 4, 6. | At baseline (week 0) and at week 6 (for part I of study) and week 4 (part II of study)
  The beliefs about consequences scale has not yet been validated but has been adapted from previous research on beliefs about capabilities by Wallin, Boström and Gustavsson (2012). The scale is a 5-point sale from 1- not at all to 5- extremely. Higher scores indicate higher beliefs about consequences.
Change in body weight from baseline to week 4,6 | Baseline(week 0) and at week 6 (for part I of study) and week 4 (part II of study)
  Self-reported weight (in kg/lbs) collected at baseline and at week 6 (for part I of study) and week 4 (part II of study)

OTHER OUTCOMES:
Personality traits on a BFI-2S questionnaire at baseline | At baseline (week 0)
  The BFI-2S questionnaire (Soto and John, 2017) is a validated questionnaire to assess the Big Five Personality domains of an individual.
Level of need for autonomy on the nutrition causality orientation scale at baseline. | At baseline (week 0)
  The nutrition causality orientation scale is a measure of the need for autonomy in nutrition-related decisions. It is not yet validated but is adapted from previous research on the validated health causality orientation scale (Smit and Bol, 2020). The scale is a 7-point scale, with 1 being strongly disagree to 7 being strongly agree.

CONTACTS AND LOCATIONS:
Locations (1):
- Liverpool John Moores University, Liverpool, United Kingdom

IPD SHARING:
Plan to Share IPD: No
The deidentified individual participant data may be shared with other researchers on a case by case basis upon request and subject to Data Protection Officer approval.

REFERENCES:
- [Background] Impey SG, Hearris MA, Hammond KM, Bartlett JD, Louis J, Close GL, Morton JP. Fuel for the Work Required: A Theoretical Framework for Carbohydrate Periodization and the Glycogen Threshold Hypothesis. Sports Med. 2018 May;48(5):1031-1048. doi: 10.1007/s40279-018-0867-7. PMID 29453741
- [Background] Dunne DM, Lefevre C, Cunniffe B, Tod D, Close GL, Morton JP, Murphy R. Performance Nutrition in the digital era - An exploratory study into the use of social media by sports nutritionists. J Sports Sci. 2019 Nov;37(21):2467-2474. doi: 10.1080/02640414.2019.1642052. Epub 2019 Jul 26. PMID 31345110
- [Background] Yan X, Ghosh P, Chakraborty B. Sample size calculation based on precision for pilot sequential multiple assignment randomized trial (SMART). Biom J. 2021 Feb;63(2):247-271. doi: 10.1002/bimj.201900364. Epub 2020 Jun 11. PMID 32529788
- [Background] Bentley MRN, Mitchell N, Backhouse SH. Sports nutrition interventions: A systematic review of behavioural strategies used to promote dietary behaviour change in athletes. Appetite. 2020 Jul 1;150:104645. doi: 10.1016/j.appet.2020.104645. Epub 2020 Feb 27. PMID 32112958
- [Background] Heikura IA, Stellingwerff T, Burke LM. Self-Reported Periodization of Nutrition in Elite Female and Male Runners and Race Walkers. Front Physiol. 2018 Dec 3;9:1732. doi: 10.3389/fphys.2018.01732. eCollection 2018. PMID 30559680
- [Background] Heikura IA, Burke LM, Mero AA, Uusitalo ALT, Stellingwerff T. Dietary Microperiodization in Elite Female and Male Runners and Race Walkers During a Block of High Intensity Precompetition Training. Int J Sport Nutr Exerc Metab. 2017 Aug;27(4):297-304. doi: 10.1123/ijsnem.2016-0317. Epub 2017 Apr 7. PMID 28387576
- [Background] Mazorra Blanco, Rodrigo; (2019) A Data Science approach to behavioural change: large scale interventions on physical activity and weight loss. Doctoral thesis (Ph.D), UCL (University College London).
- [Background] Soto CJ, John OP. Short and extra-short forms of the Big Five Inventory-2: The BFI-2-S and BFI-2-XS. Journal of Research in Personality. 2017; 68:69-81.
- [Background] Stich C, Knauper B, Tint A. A scenario-based dieting self-efficacy scale: the DIET-SE. Assessment. 2009 Mar;16(1):16-30. doi: 10.1177/1073191108322000. Epub 2008 Aug 14. PMID 18703821
- [Background] Smit ES and Bol N. From self-reliers to expert-dependents: identifying classes based on health-related need for autonomy and need for external control among mobile users. Media Psychology. 2020; 23(3): 391-414.
- [Background] Wallin L, Bostrom AM, Gustavsson JP. Capability beliefs regarding evidence-based practice are associated with application of EBP and research use: validation of a new measure. Worldviews Evid Based Nurs. 2012 Aug;9(3):139-48. doi: 10.1111/j.1741-6787.2012.00248.x. Epub 2012 Mar 27. PMID 22458331